CLINICAL TRIAL: NCT01173042
Title: Pilot Study of the Effect of Peanut Consumption on Postprandial Inflammatory Status, Glucose and Triglycerides
Brief Title: Effects of Peanut Consumption on Postprandial Inflammation, Glucose and Triglycerides
Acronym: PKEPEANUT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: The Peanut Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PKE105
Record Dates: First submitted 2010-04-13; First posted 2010-07-30 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
Keywords: Overweight; Obese
MeSH Terms: conditions — Cardiovascular Diseases; Overweight; Obesity | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Shake containing heavy whipping cream, glucose and chocolate syrup
  Interventions: Dietary Supplement: Glucose and whipping cream
- Peanut (Experimental): Shake containing control (whipping cream, glucose and chocolate syrup) + 3oz of peanuts
  Interventions: Dietary Supplement: Peanuts
- Oil blend (Experimental): Shake containing control (heavy whipping cream, glucose and chocolate syrup) + oil blend (equivalent to fatty acids provided in 3oz peanuts)
  Interventions: Dietary Supplement: Oil Blend

INTERVENTIONS:
Dietary Supplement: Peanuts — Shake containing 3.0oz of peanuts (including skin) + control (heavy whipping cream, glucose and chocolate syrup)
  Arms: Peanut
Dietary Supplement: Glucose and whipping cream — An oral liquid glucose (75g) and fat (high saturated fat from 60g heavy whipping cream) load. Chocolate syrup is added for flavor.
  Arms: Control
Dietary Supplement: Oil Blend — Shake containing an oil blend (sunflower, sesame, olive and palm oils) + control (heavy whipping cream, glucose and chocolate syrup). The amount of oil added to the control will provide an equivalent amount of fat to that provided in 3 oz (85g) of peanuts
  Arms: Oil blend

SUMMARY:
This pilot study will investigate the effects of acute peanut consumption on markers of inflammation, triglycerides and glucose. The hypothesis is that a high glucose/SFA meal will increase postprandial production of the inflammatory marker, C-reactive protein (CRP), and that the addition of peanuts to the control meal will reduce the production of CRP, as well as triglycerides and glucose.

DETAILED DESCRIPTION:
Previous research has demonstrated that a single meal high in saturated fatty acids (SFA) and glucose can induce increases in IL-6, TNF-α and CRP in abdominally obese and diabetic subjects. As over two-thirds of the U.S. population is overweight or obese, it is important to identify foods that can attenuate postprandial increases in lipids, glucose and inflammation in this population. Therefore, the purpose of the pilot study is to determine whether a high SFA / high glucose control meal will induce an acute inflammatory response in overweight individuals, and whether the addition of peanuts to this meal will ameliorate this response. To ensure that these effects are due to peanuts, and not to the increase in total fat, we will compare this response to another test meal that includes an oil blend with a similar fatty acid composition to peanuts.

ELIGIBILITY:
Inclusion Criteria:

* BMI >28
* LDL_C below 130 mg/dl
* TG below 350 mg/dl
* Blood pressure within normal ranges (below 140/90 mmHg)

Exclusion Criteria:

* Smoking
* Allergies to peanuts or dairy products
* Known intolerance for high fat meals
* History of CVD, kidney disease, diabetes or inflammatory disease
* Use of non-steroidal anti-inflammatories or immunosuppressants
* Conditions requiring the use of steroids
* Use of medication or supplements for elevated lipids, blood pressure or glucose

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Serum C-reactive protein | 0min
Serum C-reactive protein | 60 min
Serum C-reactive protein | 120 min
Serum C-reactive protein | 240 min

SECONDARY OUTCOMES:
Serum Glucose | 0 min
Serum Insulin | 0 min
Serum Triglycerides | 0 min
Serum Glucose | 60 min
Serum Glucose | 120 min
Serum Glucose | 240 min
Serum Insulin | 60 min
Serum Insulin | 120 min
Serum Insulin | 240 min
Serum Triglycerides | 60 min
Serum Triglycerides | 120 min
Serum Triglycerides | 240 min

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Hill, Ph.D, Principal Investigator — Penn State University, Department of Nutritiontal Sciences; Penny M. Kris-Etherton, Ph.D, Principal Investigator — Penn State University, Department of Nutritional Sciences; Li Wang, Study Director — Penn State University, Department of Nutritional Sciences
Locations (1):
- Penn State University, University Park, Pennsylvania, United States